CLINICAL TRIAL: NCT03644069
Title: A Phase 2 Randomized, Double-blind, Placebo-controlled Study in HLA-DQ2.5+ Adults With Celiac Disease to Assess the Effect of Nexvax2 on Symptoms After Masked Gluten Food Challenge
Brief Title: A Study of the Safety, Efficacy and Tolerability of Nexvax-2 in Patients With Celiac Disease (CeD)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ImmusanT, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Nexvax2-2006
Record Dates: First submitted 2018-05-21; First posted 2018-08-23 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Celiac Disease; Celiac; Intestinal Disease; Malabsorption Syndromes; Gastrointestinal Disease; Digestive System Disease; Gluten Sensitivity; Autoimmune Diseases
MeSH Terms: conditions — Celiac Disease; Intestinal Diseases; Malabsorption Syndromes; Gastrointestinal Diseases; Digestive System Diseases; Autoimmune Diseases | interventions — Nexvax2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nexvax2 (Experimental)
  Interventions: Biological: Nexvax2
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Nexvax2 — Nexvax2 subcutaenous (SQ) injections: 32 in total, at twice weekly intervals
  Arms: Nexvax2
Biological: Placebo — Placebo SQ injections: 32 in total, at twice weekly intervals
  Arms: Placebo

SUMMARY:
A randomized, double-blind, placebo-controlled clinical study in human leukocyte antigen (HLA)-DQ 2.5+ adults with celiac disease (CeD).

DETAILED DESCRIPTION:
A phase 2, randomized, double-blind, placebo-controlled clinical study of Nexvax2, in adults subjects with confirmed CeD who have been following a gluten free diet for at least 12 consecutive months prior to screening. This study will evaluate efficacy of Nexvax2 administered subcutaneously. The study plan consists of 3 periods: a screening period of 6 weeks, an approximately 16 week treatment period, and a 4 week post-treatment observational follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 to 70 years of age (inclusive)
* History of medically diagnosed celiac disease (CeD) that included duodenal biopsy
* Maintenance of gluten free diet (GFD) for at least 12 consecutive months prior to screening.
* Willingness to consume a moderate amount of gluten
* Able to read and understand English
* Worsening of GI symptoms in response to an oral gluten challenge
* HLA DQ 2.5 positive

Exclusion Criteria:

* Unwilling or unable to perform self-injections
* History of inflammatory bowel disease and/or microscopic colitis.
* Any medical condition or lab abnormality that in the opinion of the investigator may interfere with study conduct or would impact the immune response (other than CeD), confound interpretation of study results, or pose an increased risk to the subject.
* Use of immunomodulatory or immune-suppressing medical treatment during the 6 months prior to screening
* Use of oral or parenteral immunomodulatory corticosteroids, within the 6 weeks prior to screening. Topical or inhaled corticosteroids are acceptable.
* Receipt of any investigational drug or participation in another clinical study within 6 months prior to screening.
* Females who are lactating or pregnant
* Receipt of any vaccine within 1 week prior to planned first day of the treatment period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Nexvax2 compared to placebo in reducing Celiac Disease (CeD) associated GI symptoms. | 79 to 93 days after baseline
  Measured by the CeD Patient Reported Outcome (CeD PRO) between baseline and day of the first masked food challenge (MFC) containing gluten. The CeD PRO captures patient ratings for a number of CeD-associated symptoms, on a 0 to 10 scale, with 0 being absent or no symptoms, and 10 being the most severe symptoms. The Total GI domain score is calculated as an average of summed average and individual symptom scores relevant to the GI tract, to yield a value of 0 to 10.

SECONDARY OUTCOMES:
Evaluate efficacy of Nexvax 2 compared with placebo on immune-system activation after the first MFC containing gluten. | 79 to 93 days after baseline
  Differences in levels of pharmacodynamic markers between baseline and day of the first MFC containing gluten.
Evaluate efficacy of Nexvax2 compared with placebo in reducing CeD associated GI symptom sub-domains. | 79 to 93 days after baseline
  Differences in daily GI symptom domain score between baseline and day of the first MFC containing gluten.
Evaluate efficacy of Nexvax2 compared with placebo in reducing individual GI symptoms. | 79 to 93 days after baseline
  Differences in each of the individual GI item scores in the CeD PRO between baseline and day of the first MFC containing gluten. GI symptoms assessed on the CeD PRO include abdominal cramping, abdominal pain, bloating, diarrhea, gas, loose stool, and nausea. Each are rated on a 0 to 10 scale, where 0 is absent and 10 is the most severe.
Incidence of Treatment-Emergent Adverse Events (TEAEs) in assessing safety and tolerability of Nexvax2. | Study Duration: 21 weeks
  Treatment emergent adverse events (TEAEs) will be summarized by treatment arm, severity, relationship to study drug and to known or potential gluten exposure, and phase of treatment and presented as the number and percentage of patients reporting an event(s) as well as the number of events reported.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Anderson, PhD, FRACP, Study Chair — ImmusanT, Inc.
Locations (41):
- United States (28):
  - Diablo Clinical Research, Walnut Creek, California
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Alliance Medical Research, Lighthouse PT, Florida
  - Grand Teton Research Group, Idaho Falls, Idaho
  - UCMC - Center for Clinical Cancer Genetics and Global Health, Chicago, Illinois
  - PMG Research of McFarland Clinic, Ames, Iowa
  - University of Iowa, Iowa City, Iowa
  - Heartland Research Associates, Wichita, Kansas
  - Clinical Research Institute of Michigan, Chesterfield, Michigan
  - Center for Digestive Health, Troy, Michigan
  - West Michigan Clinical Research Center, Wyoming, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - AB Clinical Trials, Las Vegas, Nevada
  - ActivMed Practices & Research, Portsmouth, New Hampshire
  - Long Island Gastrointestinal Research Group, Great Neck, New York
  - Drug Trials America, Hartsdale, New York
  - Celiac Disease Center at Columbia University, New York, New York
  - PMG Research of Piedmont Healthcare, Statesville, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Great Lakes Gastroenterology Research, Mentor, Ohio
  - Thomas Jefferson University Hospitals - Center City Campus, Philadelphia, Pennsylvania
  - Ocean State Clinical Research Partners, Lincoln, Rhode Island
  - Omega Medical Research, Warwick, Rhode Island
  - Coastal Carolina Research, Mt. Pleasant, South Carolina
  - Digestive Health Research, Hermitage, Tennessee
  - Texas Digestive Disease Consultants, Southlake, Texas
  - Advanced Research Institute, South Ogden, Utah
  - Allegiance Research Specialists, Wauwatosa, Wisconsin
- Australia (9):
  - The Wesley Hospital - The Wesley Research Institute, Auchenflower, Queensland
  - Coral Sea Clinical Research Institute, Mackay, Queensland
  - Clinical Trials Centre - University of the Sunshine Coast, Sippy Downs, Queensland
  - The University of Queensland - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, Southern Australia
  - Eastern Health-Box Hill Hospital, Box Hill, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - The Royal Melbourne Hospital - The Walter and Eliza Hall Institute of Medical Research, Parkville, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- New Zealand (4):
  - Auckland Clinical Studies, Auckland
  - Gastroenterology and Endoscopy Specialists, Christchurch
  - P3 Research Limited, Havelock North
  - P3 Research Limited, Mount Cook

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tye-Din JA, Daveson AJM, Goel G, Goldstein KE, Hand HL, Neff KM, Popp A, Taavela J, Maki M, Isola J, Williams LJ, Truitt KE, Anderson RP; RESET CeD Study Group. Efficacy and safety of gluten peptide-based antigen-specific immunotherapy (Nexvax2) in adults with coeliac disease after bolus exposure to gluten (RESET CeD): an interim analysis of a terminated randomised, double-blind, placebo-controlled phase 2 study. Lancet Gastroenterol Hepatol. 2023 May;8(5):446-457. doi: 10.1016/S2468-1253(22)00428-9. Epub 2023 Mar 7. PMID 36898393
- [Derived] Tye-Din JA, Daveson AJM, Goldstein KE, Hand HL, Neff KM, Goel G, Williams LJ, Truitt KE, Anderson RP; RESET CeD Study Group. Patient factors influencing acute gluten reactions and cytokine release in treated coeliac disease. BMC Med. 2020 Nov 26;18(1):362. doi: 10.1186/s12916-020-01828-y. PMID 33239013
- See also: ImmusanT — http://www.immusant.com/